CLINICAL TRIAL: NCT06067464
Title: Evaluation of Peripheral Pulse-oximeter Derived Perfusion Index as a Prognostication Tool for High Quality Cardiopulmonary Resuscitation and Return of Spontaneous Circulation
Brief Title: Evaluation of Perfusion Index as a Prognostication Tool for High Quality Cardiopulmonary Resuscitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, ICU, fellow of intensive care medicine, National Hepatology & Tropical Medicine Research Institute
Other Study IDs: 28-2023
Record Dates: First submitted 2023-08-28; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In order to monitor and improve cardiopulmonary resuscitation(CPR) quality, there is need for tools that provide real time feedback to responders. The use of invasive arterial pressure monitoring and end tidal carbon dioxide (ETCO2) as quality measures of CPR. Invasive pressure measurements are timeconsuming and cumbersome in resuscitation situations, and are very rarely practical. ETCO2 measurements require presence of a capnometer with an advanced airway.

High quality chest compression will result inETCO2 between 2-2.5KPa. A rapid increase in ETCO2 on waveform capnography may enable ROSC to be detected while continuing chest compression and can be used as a tool to withhold the next dose of bolus adrenaline injection.

Pulse oximetry, which noninvasively detects the blood flow of peripheral tissue, has achieved widespread clinical use. It was noticed that the pulse waveform frequency can reflect the rate and interruption time of chest compression(CC) during cardiopulmonary resuscitation(CPR).

The perfusion index (PI) is obtained from pulse oximetry and is computed as the ratio of the pulsatile (alternating current) signal to the non-pulsatile (direct current) signal of infra-red light, expressed as a percentage;PI =ACIR/DCIR∗100% (i.e. AC = pulsatile component of the signal, DC = non-pulsatile component of the signal, IR = infrared light).

PI shows the perfusion status of the tissue in the applied area for an instant and a certain time interval. The PI value ranges from 0.02% (very weak) to 20% (strong).Peripheral PI has been proposed for different clinical uses with some applications in critical patients.

The purpose of this study is to evaluate the role of pulse-oximeter derived perfusion index for high quality CPR and as aprognostication tool of ROSC during in-hospital cardiac arrest in comparison to ETCO2 reading.

DETAILED DESCRIPTION:
After approval by NHTMRI-IRB Ethical Committee.All demographic data will be obtained including the patients' age, sex, associated co-morbidities (e.g. diabetes mellitus & hypertension), cause of cardiac arrest, and duration of CPR.

Resuscitation for patients will be held according to ERC (Advanced life support) ALS Algorithm 2021.1 Electrocardiogram of manual defibrillator, pulse oximeter (Nihon-Kohden, Mindray) will be attached to the middle finger or thumb7 and the capnography will be attached between endotracheal tube and Bag mask valve. Both readings of the ETCO2 and pulse oximeter derived perfusion index will be recorded every minute till the end of CPR.The medical staff did not alter the patient's treatment based on PI results. One week and 30 day survival will be followed.

ELIGIBILITY:
Inclusion Criteria:

* The subjects are adults aged between 18 & 75years who developed in-hospital cardiac arrest and cardiopulmonary resuscitation for at least 3 minutes either in emergency departments or wards or Intensive care units in the National Hepatology and Tropical Medicine Research Institute (NHTMRI) and Alexandria University

Exclusion Criteria:

* Patients will be excluded from the study ifpregnant,known peripheral vascular disease or >2 vasopressors with the maximum doses or in the presence of nail polish as readings from pulse oximeter will be distorted .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Resuscitation for patients will be held according to ERC (Advanced life support) ALS Algorithm 2021.1 Electrocardiogram of manual defibrillator, pulse oximeter (Nihon-Kohden, Mindray) will be attached to the middle finger or thumb7 and the capnography will be attached between endotracheal tube and Bag mask valve. Both readings of the ETCO2 and pulse oximeter derived perfusion index will be recorded every minute till the end of CPR.The medical staff did not alter the patient's treatment based on PI results. One week and 30 day survival will be followed.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
prognostication | during 20 minutes of CPR
  evaluate the role of PI as a prognostic tool for high quality CPR in comparison with ETCO2.

SECONDARY OUTCOMES:
prognostication | during20 minutes of CPR
  of PI as a prognostication tool for ROSCin comparison to the readings of ETCO2
survival | one week and 30 days
  either higher PI during CPR associated with one week and 30 day survival

CONTACTS AND LOCATIONS:
Locations (1):
- NHTMRI, Cairo, Egypt